CLINICAL TRIAL: NCT06296992
Title: Type 1 Diabetes, Exercise and Mentoring (TEAM) Trial: A Randomized Controlled Pilot Trial Using Peer Mentorship to Increase Physical Activity and Quality of Life in Adolescents With Type 1 Diabetes
Brief Title: Type 1 Diabetes, Exercise and Mentoring Trial
Acronym: TEAM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Jon McGavock, Professor, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: B2023:035
Record Dates: First submitted 2024-01-15; First posted 2024-03-06 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Type 1 Diabetes; Physical Activity
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 12-week TEAM peer mentor program (Experimental): A 12-week peer-led behavioural intervention that supports increased physical activity. It will consist of 3 weekly contacts between participants and peer mentors that will be a mix of in-person, virtual, and texting. The intervention components and communication between adolescents and peer mentors with T1D will be guided by SDT, and designed to overcome the key psychosocial barriers to PA. The peer mentors that complete the training will deliver a 12-week intervention to increase behavioural skills that foster autonomy for goal setting and overcoming barriers to PA.
  Interventions: Behavioral: 12-week TEAM peer mentor program
- 12-week waitlist control (No Intervention): A 12-week waitlist control group that receives usual care, including standard educational resources developed by the Canadian Society of Exercise Physiology for adopting and sustaining daily PA. Adolescents randomized to the control arm will be offered the 12 week intervention following the 24 week follow-up time point.

INTERVENTIONS:
Behavioral: 12-week TEAM peer mentor program — A 12-week peer-led behavioural intervention that supports increased physical activity. It will consist of 3 weekly contacts between participants and peer mentors that will be a mix of in-person, virtual, and texting. The intervention components and communication between adolescents and peer mentors with T1D will be guided by SDT, and designed to overcome the key psychosocial barriers to PA. The peer mentors that complete the training will deliver a 12-week intervention to increase behavioural skills that foster autonomy for goal setting and overcoming barriers to PA.
  Arms: 12-week TEAM peer mentor program

SUMMARY:
The proposed study aims to improve the psychosocial health of adolescents living with type 1 diabetes (T1D). The study will generate knowledge and support knowledge mobilization about the effectiveness of a novel model of care for psychosocial health and self-management for adolescents living with type 1 diabetes (T1D). The novel model of care is the recruitment and training if young adult mentors to deliver a behavioural intervention that empowers adolescents with T1D to increase daily physical activity. The study will also advance the development and implementation of this peer mentoring model to improve the psychosocial health of adolescents with T1D.

DETAILED DESCRIPTION:
Rationale: Empowering adolescents with type 1 diabetes (T1D) to increase daily physical activity (a cornerstone behaviour in diabetes self-management) is well-defined knowledge gap in pediatric endocrinology clinical practice. Adopting a lifestyle that includes regular physical activity (PA) is essential for the optimal health and quality of life (QoL) of adolescents living with T1D, however Diabetes Canada clinical practice guidelines provide no evidence for optimal behavioural approaches for achieving the extensive self-management behaviours needed to prevent diabetes-related complications during a critical stage of psychological, social and emotional development. As such, daily PA levels remain low in adolescents with T1D and many do not meet current recommendations for daily PA. The aim of this pilot trial is to assess the feasibility, preliminary efficacy and safety of a novel peer-led behavioural intervention to increase PA and quality of life for adolescents living with T1D.

Methodology: Investigators will conduct a pilot randomized controlled trial comparing a peer-led, behavioural intervention, to standard of care on daily PA and quality of life. Investigators will also conduct a qualitative study within the trial to understand the contextual factors that influenced the peer mentoring approach to empowering adolescents with T1D.

Population: Sixty adolescents 13-17 years of age living with T1D from 2 sites in Canada who will be randomized 2:1 to intervention or control arms, respectively.

Intervention Arm: A 12-week behavioural intervention guided by the tenets of self-determination theory, and led by a physically active young adult mentors, 21-30 yrs of age living with T1D. Mentors will rely on motivational interviewing skills to support adolescents living with T1D to increase daily PA by fostering a sense of autonomy for goal setting and self-management skill acquisition, competency in their ability to increase daily PA without compromising glucose management and a sense of relatedness to a community of adolescents overcoming similar challenges.

Control Arm: Adolescents in the wait-list control arm will receive standard clinical recommendations to increase daily PA.

Investigators will also conduct a qualitative study with 10 adolescents who participated in the intervention. The qualitative component will attempt to (1) identify the complex factors that influenced adherence to the intervention; (2) determine the appropriateness and relevance of peer mentoring for adolescents with T1D; (3) explore sex, gender and psychosocial-specific factors related to the delivery of the peer mentoring intervention; and (4) explore possible novel mediators of the effect of the study arms on psychosocial health, quality of life and health behaviours.

Timing: Feasibility and fidelity outcomes will be assessed throughout the trial and at the 12-week time point.

Patient-engagement: Patient co-researchers from Canada and Ireland participated in several formative studies that informed this proposal. They co-designed the novel peer-led intervention and all aspects of the trial outlined in this proposal.

Importance: The results of this trial will inform a larger trial to provide much needed empirical evidence for inform pediatric diabetes clinical practice guidelines for behavioural strategies to improve self management and quality of life for adolescents living with T1D.

ELIGIBILITY:
Inclusion Criteria:

* want to increase their daily PA
* currently use a continuous glucose monitor (CGM)

Exclusion Criteria:

* were diagnosed with T1D within 12 months of randomization
* have diabetes secondary to medications or surgery
* have cancer
* evidence of drug/alcohol abuse
* have an eating disorder
* an orthopedic injury or illness that would limit their ability to engage in daily PA
* a suicide attempt in the previous 12 months
* are pregnant

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Enrollment rates | during the study period of approximately three years.
  Defined as the number of (i) adolescents who consent to participate and are randomized to one of the two study arms during the study period of approximately three years and (ii) the number of young adults who agree and complete the training to become peer mentors to the adolescents during the study period of approximately three years.
Adherence to the intervention arms | during the study period of approximately three years
  Defined as the percentage of prescribed sessions that adolescents attended during the trial period of approximately three years
Retention for follow-up measurements | during the study period of approximately three years.
  Defined as the percentage of adolescents who complete follow-up measurements during the study period of approximately three years.

SECONDARY OUTCOMES:
Physical activity | Baseline, week 12, week 24
  Daily moderate to vigorous physical activity measured for seven days with a waist mounted accelerometer
Quality of Life (DQOL) | Baseline, week 12, week 24
  The Health-Related Quality of Life in persons living with diabetes (DQOL) will be used to measure overall quality of life. Lower scores indicate better quality of life.
Quality of Life (PedsQL 4.0) | Baseline, week 12, week 24
  Quality of Life (PedsQL 4.0) will be used to measure the condition-specific quality of life. Lower scores indicate better quality of life.

OTHER OUTCOMES:
Diabetes Distress | Baseline, week 12, week 24
  The Problem Areas in Diabetes-Teen (PAID-peds) survey has the best psychometric properties for adolescents and young adults. With the PAID-T, adolescents use a 6-point scale (1 -not a problem to 6 -a serious problem) to rate various sources of distress over the past month.
Mastery | Baseline, week 12, week 24
  The Perceived Competence for Diabetes Scale (PCDS) assesses the degree to which people with diabetes feel they can manage the everyday aspects of diabetes care. The PCDS contains four statements, rated on a 7-point Likert scale, with higher scores representing better respondent performance.
Autonomy | Baseline, week 12, week 24
  The Treatment Self-Regulation Questionnaire (TSRQ) is a theoretically derived scale that assesses the degree of autonomous self-regulation regarding why people engage or would engage in healthy behavior and is designed to assess the different forms of motivation within SDT.
Motivation for physical activity (LCE) | Baseline, week 12, week 24
  The Locus of Causality for Exercise Scale (LCE) is a brief, three-item scale designed to assess the extent to which individuals feel that they freely choose to exercise rather than feeling that they have to for an external reason (i.e. parents/external expectations). Higher scores indicate higher self-determination.
Readiness for change | Baseline, week 12, week 24
  Readiness for change will be assessed using the PA counselling readiness questionnaire (PACE).
Motivation to engage in exercise | Baseline, week 12, week 24
  The Behavioral Regulation in Exercise Questionnaire-3 (BREQ3) is a measure of motivation to engage in exercise from an SDT perspective.
Motivation for Physical Activity (EMI-2) | Baseline, week 12, week 24
  The Exercise Motivations Inventory-2 (EMI-2) examines the significance of exercise motives from the perspective of self-determination theory.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan McGavock, Principal Investigator — University of Manitoba / the Children's Hospital Research Institute of Manitoba
Locations (2):
- Canada (2):
  - the Children's Hospital Research Institute of Manitoba and the University of Manitoba, Winnipeg, Manitoba
  - Trillium Health Partners, Mississauga, Ontario

IPD SHARING:
Plan to Share IPD: No